CLINICAL TRIAL: NCT04755218
Title: A Cluster Randomized Trial of Labor Induction With Oral Versus Vaginal Misoprostol
Brief Title: Labor Induction With Oral Versus Vaginal Misoprostol
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Emily Adhikari, Principal Investigator, University of Texas Southwestern Medical Center
Other Study IDs: STU 2020-1395
Record Dates: First submitted 2021-02-05; First posted 2021-02-16 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Pregnancy; Labor, Induced
Keywords: Pregnancy; Labor induction; Cervical Ripening; misoprostol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaginal Misoprostol: Patients will receive vaginal misoprostol 25 micrograms given every 3 hours for a maximum of 5 doses. Although labeled "experimental" for comparison purposes, this is not an experimental intervention, as the method is a currently accepted standard of care for cervical ripening and labor induction in the United States
- Oral Misoprostol: Patients will receive standard oral misoprostol 100 micrograms given every 4 hours for a maximum of 2 doses according to current labor induction protocol

SUMMARY:
This study will compare vaginal and oral misoprostol, to determine whether a vaginal misoprostol regimen achieves a higher vaginal delivery rate in a real-world, high-volume setting, and whether this regimen reduces time and oxytocin need on a high-volume Labor and Delivery unit at Parkland Hospital.

Our primary hypothesis is that among women with singleton, term pregnancies, cervical dilation 2cm or less, and indicated labor induction, the rate of vaginal delivery is significantly increased when a standardized vaginal misoprostol regimen is used, compared with a standardized oral misoprostol regimen.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the use of a standardized vaginal misoprostol regimen will result in a decreased primary cesarean delivery rate among women with a cervical dilation of 2 centimeters of less who require induction of labor at term, compared with the currently used oral misoprostol regimen. We also aim to evaluate oxytocin use, time to delivery, uterine activity, indication for cesarean delivery, intrapartum and postpartum infectious morbidities, excess blood loss at delivery, and adverse neonatal outcomes in the overall population as well as nulliparous women specifically.

This will be a prospective, cluster-randomized clinical trial to compare the rate of vaginal delivery achieved when two standards of care are used across a large population of women with indication for labor induction at Parkland Hospital. Eligible participants will include nulliparous and multiparous women at 37 weeks gestation or greater, with a living, singleton fetus and no major fetal malformations, in cephalic presentation, with intact membranes, no prior uterine scar, who qualify for prostaglandin administration and who have a cervical dilation of 2 centimeters or less, measured at the level of the internal os. Patients with non-reassuring fetal status, active herpes outbreak, a prior uterine scar, or any contraindication to prostaglandins (including 4 or more painful contractions per 10 minutes prior to prostaglandin administration) will be excluded from participation in the study.

Computer-generated cluster randomization will occur on a weekly basis for all study participants, to either the vaginal misoprostol regimen (study group) or to oral misoprostol regimen (control group).

According to the randomization protocol each week, participants will be randomized to either the oral misoprostol standard of care (control group) or vaginal misoprostol standard of care (study group). The study group will receive vaginal misoprostol 25 mcg every 3 hours for a maximum of 5 doses in those who meet criteria for prostaglandin administration. The control group will receive oral misoprostol 100 micrograms given every 4 hours for a maximum of 2 doses. Misoprostol will not be administered to patients who have progressed to active labor, defined as 4 centimeters cervical dilation. Intravenous oxytocin will be administered according to current PHHS protocol for both groups.

No direct contact between the research team and patients will be required, as this is a systematic comparison of two standards of care.

The primary outcome will be the rate of vaginal delivery.

Secondary outcomes will include maternal and neonatal outcomes.

Maternal outcomes will include time to delivery, time (hours) of oxytocin, need for oxytocin, indication for cesarean delivery, labor analgesia, clinical chorioamnionitis, tachysystole, hyperstimulation syndrome, excess estimated blood loss, transfusion at delivery, endometritis, surgical site infection, uterine rupture, and unplanned hysterectomy.

Neonatal outcomes will include meconium-stained amniotic fluid, umbilical cord pH <7.0, 5-minute Apgar <4, neonatal intubation or ventilation in the delivery room, neonatal sepsis, and neonatal intensive care (NICU) admission.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous and multiparous pregnant women
* 37 weeks gestation or greater
* Living, singleton fetus
* No major fetal malformations
* Cephalic presentation
* No prior uterine scar
* Intact fetal membranes
* Qualifies for prostaglandin administration according to current Parkland protocol
* Have a cervical dilation of 2 centimeters or less, measured at the level of the internal os
* Have an indication for induction or attempted induction of labor according to Parkland protocol

Exclusion Criteria:

* Non-reassuring fetal status
* Active herpes outbreak
* Prior uterine scar
* Contraindication to prostaglandins according to current Parkland protocol (including 4 or more painful contractions per 10 min prior to prostaglandin administration)
* Contraindication to vaginal delivery

Min Age: 10 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nulliparous and multiparous pregnant women at 37 weeks gestation or greater, with a living, singleton fetus and no major fetal malformations, in cephalic presentation, no prior uterine scar, with intact fetal membranes, who qualify for prostaglandin administration and who have a cervical dilation of 2 centimeters or less, measured at the level of the internal os, requiring induction at Parkland Health and Hospital System.
Sampling Method: Probability Sample
Enrollment: 2546 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-09-18 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Vaginal Delivery | at delivery
  vaginal delivery at first induction

SECONDARY OUTCOMES:
Time to Delivery | from start of induction agent to time of delivery
  time (in hours) from start of induction agent to delivery at first induction
Time (hours) of Oxytocin | at delivery
  time (in hours) from start of Oxytocin until turned off for delivery
Need for Oxytocin | at delivery
  administration of Oxytocin to facilitate labor contractions
Indication for Cesarean Delivery | at delivery
  among women delivered by cesarean, the indication for cesarean
Use of Epidural During Labor | at delivery
  use of epidural between the start of induction and delivery
Presence of Chorioamnionitis | at delivery
  intrapartum fever (temp greater than or equal to 38 degrees C) with clinical concern for infection and no other identified cause
Number of Participants with Uterine Hyperstimulation Syndrome | at delivery
  tachysystole accompanied by fetal heart rate decelerations
Number of Participants with Excess Blood Loss | at delivery
  Maternal excess blood loss is defined as >500mL for vaginal and >1000mL for cesarean delivery
Number of Participants with Blood Transfusion | at delivery
  administration of blood products related to delivery blood loss
Number of Participants with Puerperal Fever and/or Endometritis | immediately after delivery to discharge from the hospital, or up to 4 weeks postpartum
  maternal fever recorded in the time after delivery, but prior to discharge from the hospital, with or without clinical assessment of endometritis
Surgical Site Infection | from time of birth until the time of discharge, or up to 4 weeks postpartum
  documentation of cellulitis, organisms grown on wound culture, or superficial or deep space surgical site infection with or without purulent drainage requiring readmission
Number of Participants with Uterine Rupture | at delivery
  spontaneous separation of myometrium in a previously intact, unscarred uterus
Number of Participants with Unplanned Hysterectomy | immediately after delivery to discharge from the hospital, or up to 4 weeks postpartum
  unplanned removal of the uterus following delivery of the fetus
Number of Participants with Meconium-Stained Amniotic Fluid | at the time of rupture of membranes or at delivery
  identification of any meconium (green tinge) in the amniotic fluid before or during delivery by a healthcare provider's assessment of gross fluid color
Number of Participants with Umbilical pH <7.0 | at delivery
  arterial or venous cord blood pH defined as < 7.0
Number of Participants with a 5-minute Apgar Score Less Than 4 | 5 minutes after time of birth
  Appearance, Pulse, Grimace, Activity, Respirations-scored from 0-2 for each component, added to make a total score and used as an assessment of initial response to newborn resuscitation, lower scores associated with poor outcomes. Here defined as Apgar <4 at 5 minutes
Number of Participants That Needed Mechanical Ventilation in Delivery Room (Yes/No) | at delivery
  intubation with mechanical support or control of neonatal breathing in the delivery room
Number of Participants with Neonatal Sepsis | from time of birth until time of discharge or up to 7 days of life, whichever comes first
  neonatal bacteremia as defined by bacterial growth in blood cultures
Number of Participants with NICU Admission Order | from time of birth until the time of discharge or up to 7 days of life, whichever comes first.
  admission order to neonatal intensive care unit (NICU) placed between the time of delivery and infant discharge

CONTACTS AND LOCATIONS:
Overall Officials: Emily H Adhikari, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health and Hospital Systems, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adhikari EH, McGuire J, Lo J, McIntire DD, Spong CY, Nelson DB. Vaginal Compared With Oral Misoprostol Induction at Term: A Cluster Randomized Controlled Trial. Obstet Gynecol. 2024 Feb 1;143(2):256-264. doi: 10.1097/AOG.0000000000005464. Epub 2023 Nov 21. PMID 37989142